CLINICAL TRIAL: NCT03859843
Title: Efficacy and Antimicrobial Activity of Platelet Rich Plasma (PRP) in Acne Vulgaris : A Randomized Controlled Trial
Brief Title: Efficacy and Antimicrobial Activity of Platelet Rich Plasma (PRP) in Acne Vulgaris
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hiba A H alshaaby, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP in Acne Vulgaris
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Platelet-Rich Plasma; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Chemexfoliation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP (Active Comparator)
  Interventions: Combination Product: PRP
- Chemical peeling (Salycilic acid) (Active Comparator)
  Interventions: Other: Chemical peeling (Salycilic acid)
- Chemical peeling (Jessenr's solution) (Active Comparator)
  Interventions: Other: Chemical peeling (Jessener's solution)

INTERVENTIONS:
Combination Product: PRP — Ten mL of venous blood will be drawn in a syringe fill with 1.5 mL of anticoagulant solution (anticoagulant citrate dextrose solution formula A, Baxter, Deerfield, IL). The blood will be centrifuged at 160 g for 10 minutes. After the first spin, the lower red blood cell portion will be discarded, and the supernatant will be centrifuged at 400 g for 10 minutes. The resulting pellet of platelets will be mixed with 1.5 mL of supernatant, which make 1.5 mL of PRP. One mL of 3% calcium chloride will be added to the PRP to induce platelet activation.
  Arms: PRP
Other: Chemical peeling (Salycilic acid) — SA is a 2-hydroxybenzoic acid (from willow tree) used for superficial peeling due to its strong keratolytic and comedo- lytic properties. It promotes shedding of epidermal cells and due to its lipophilic properties can penetrate comedones and pores to prevent clogging and neutralize bacteria. It promotes desquamation of the upper lipophilic layers of the stratum corneum.19 These chemical properties explain its popularity and success in acne patients.It also has well- documented anti-inflammatory properties.
  Arms: Chemical peeling (Salycilic acid)
Other: Chemical peeling (Jessener's solution) — is a superficial peeling agent used as adjuvant therapy for acne. it is generally proposed to break of the hydrogen bonds of keratin (keratolysis), disruption of cell membranes (cell death) and is bactericidal.
  Arms: Chemical peeling (Jessenr's solution)

SUMMARY:
Efficacy and Antimicrobial activity of Platelet Rich Plasma (PRP) in Acne Vulgaris : A randomized controlled trial

DETAILED DESCRIPTION:
Acne vulgaris is one of the most common chronic skin diseases worldwide. The condition usually starts in adolescence, peaks at the ages of 14 to 19 years and frequently resolves by mid-twenties.

Acne is characterized by seborrhea, formation of open and closed comedones, erythematous papules and pustules and in more severe cases present with nodules, deep pustules and pseudo cysts, in many cases a degree of scarring will ensue.

Its pathophysiology includes hyperseborrhoea, abnormal follicular keratinization and Propionibacterium acnes proliferation in the pilosebaceous unit.

Acne is a significant clinical problem with sever social, psychological, and emotional implications. A mainly genetically determined host response pattern combined with bacterial ''triggering'' is generally accepted as being important for the apparently unbalanced inflammatory activity.

Acne is not an infectious disease, but three major organisms were isolated from the surface of the skin and the pilosebaceous duct of patients with acne including Propionibacterium acne, Staphylococcus epidermidis and Malassezia furfur.

Platelet rich plasma is a good choice for the treatment of acne and atrophic scars reminiscent of the course of the disease. In addition, for being autologous, it reduces the possibility of side effects, such as skin dryness and rejection.

It was demonstrated that PRP accelerates the healing process, regulates inflammation and promotes healing by inhibiting the P. acnes bacteria, additionally restoring collagen). The PRP's mechanism of action also involves the release of powerful antimicrobial peptides from the platelets' alpha granules.

Although there are few studies on the PRP's effectiveness in acne, it emerges as a potential therapeutic option in Dermatology and Aesthetic Medicine.

Due to development of resistance in microorganisms causing acne to common antibiotics and differences in species and strains of the microorganisms in different regions, this study will be undertaken to determine bacteria involve in acne vulgaris and the effect of PRP on it.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active acne vulgaris lesions (inflammatory and non-inflammatory).
* Age range from 14 to 40 years.
* Patients with any topical and systemic treatments will undergo wash out period of one month.

Exclusion Criteria:

* Patients with herpes labials, or bacterial infection; warts on the face, actinic keratosis, or skin cancer or allergy to medications.
* Systemic retinoids intake in the previous 6 months
* History of keloidal scarring.
* Patients on anticoagulant therapy or aspirin or have a coagulation issue,
* Patients with hemoglobin less than 10g\dl or platelet less than 105 micron\l
* Pregnant women
* Immunocompromised patients
* Patients with medical diseases like diabetes mellitus, epilepsy or malignancy

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2022-05-10 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 3 months
  Assess cure rate of PRP and Chemical peeling agents in treatment of Aactive Acne Vulgaris in 3 months duration and compare efficacy of all measures

IPD SHARING:
Plan to Share IPD: Undecided